CLINICAL TRIAL: NCT01010854
Title: A Phase II Study of Valproic Acid in Combination With FEC100 for Primary Therapy in Patients With Locally Advanced or Primary Metastatic Breast Cancer
Brief Title: Valproic Acid in Combination With FEC100 for Primary Therapy in Patients With Breast Cancer
Acronym: VPA-FEC100
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Premature closure for lack of efficacy.
Sponsor: University of California, San Francisco (Other)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC# 087515; NCT00437801 (obsolete NCT alias)
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; advanced; local
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VPA FEC100 (Experimental): Valproic Acid with FEC100
  Interventions: Drug: VPA FEC100

INTERVENTIONS:
Drug: VPA FEC100 — oral VPA (60 mg/kg bid) q 12h X 6 with IV 5-Fluorouracil (500 mg/m2) Epirubicin (100 mg/m2) and Cyclophosphamide (500 mg/m2)

SUMMARY:
The drugs FEC 100 (5-fluorouracil, epirubicin, and cyclophosphamide) are one of the approved options to treat Locally Advanced or Primary Metastatic Breast Cancer. In this study, the investigators will add another drug called Valproic Acid (VPA) to see whether this makes the treatment better. The addition of Valproic Acid to chemotherapy has been studied in about 65 subjects with cancer and was found to be safe and tolerable. Valproic Acid is approved by the Food and Drug Administration (FDA) for the treatment of seizures, mood swings, and migraine headaches. It is not currently approved for cancer, which is why the investigators are conducting this study.

The results of a Phase I study of Valproic Acid and FEC100 in subjects with cancer that has spread has led the investigators to believe that this combination is better than just the standard treatment alone. The investigators are now testing the combination in a study with subjects who have either a large tumor, many lymph nodes involved or patients whose tumor has spread. In addition to the treatment, a main goal of the study is to find out which subjects will benefit from this combination. In the Phase I trial the investigators noticed that while this combination appears to make the chemotherapy more effective, it did not appear to cause more side effects induced by the chemotherapy.

DETAILED DESCRIPTION:
Each year, more than 200,000 patients are diagnosed with breast cancer. While recent advances in diagnosis and treatment have rendered a large proportion of these patients curable, many patients still present with either locally advanced or metastatic breast cancer that is not amenable to potentially curative surgery. To enhance the chance of complete surgical resection of the tumor, patients with very large, locally advanced or inflammatory breast cancer will be offered neo-adjuvant therapy.

The use of systemic chemotherapy after the surgical therapy for patients with operable disease has been associated with a 25%-35% reduction in the risk of systemic relapse (Early Breast Cancer Trialists' Collaborative Group, 1998) Administration of chemotherapy prior to surgery, also referred to as neoadjuvant chemotherapy is often used in patients with inoperable, non-metastatic breast cancer. However more recently, neoadjuvant therapy has become more commonly used as it allows the direct assessment of response to systemic therapy and the collection of biological markers of therapy that are otherwise difficult to obtain. Furthermore, the relative high response rate allows the ability to surgically remove the tumor and achieve adequate tumor-free margins.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of breast cancer
* Patients must have "locally advanced" adenocarcinoma of the breast:

  * tumors > 2 cm without lymph node involvement (negative sentinel lymph node mapping)
  * tumors > 2 cm with lymph node involvement (either by positive sentinel lymph node mapping or FNA of palpable lymph node)
  * tumors of any size that show extension to the chest wall or skin, including edema, ulceration, or satellite skin nodules
  * inflammatory carcinoma (stage IIIB) that is amenable to surgery
  * tumors of any size associated with ipsilateral internal mammary nodes (stage IIIB)
  * tumors of any size associated with ipsilateral supraclavicular lymph nodes (IIIC) without other evidence of systemic metastases
  * patients may have bilateral breast cancer if both breasts are assessible for response
* Age >18 years
* Because no dosing or adverse event data are currently available on the use of VPA in combination with FEC100 in patients <18 years of age, children are excluded from this study
* ECOG performance status 0 or 1 (Karnofsky >80%)
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >3,000/mcL
  * absolute neutrophil count >1,500/mcL
  * platelets >100,000/mcL
  * total bilirubin within 1.5 x normal institutional limits
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits
* VPA has been associated with neural tube defects in the developing human fetus, for this reason and because FEC100 used in this trial are also known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Participating men must use condoms while on study and for at least 3 months after the trial has ended. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not have had any prior chemotherapy within the last 2 years
* Patients may not have been exposed to prior anthracyclines
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases are excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to VPA or FEC100.
* Patients with known congestive heart disease or LVEF fractions of <50 % (past or current), patients with known ventricular arrhythmias
* Patients taking VPA as an anti-seizure agent or for any other indications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Due to the teratogenic effects of VPA and FEC100, pregnant or lactating women are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-12-10 (Actual); Primary Completion 2010-12-12 (Actual); Study Completion 2011-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VPA FEC100
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VPA FEC100
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 56 [50 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response at Definitive Surgery
Time Frame: after 4 cycles of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | VPA FEC100
Number analyzed (Participants) | 6
Participants | 3

2. Secondary Outcome: Clinical Response Based on Tumor Measurement
Time Frame: after 4 cycles of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | VPA FEC100
Number analyzed (Participants) | 6
Participants | 3

ADVERSE EVENTS:
Arm/Group | VPA FEC100
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VPA FEC100 (N=6)
Dizziness (Nervous system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VPA FEC100 (N=6)
Hemoglobin (Blood and lymphatic system disorders) | 6
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 2
Platelets (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 6
Insomnia (General disorders) | 1
Rigors (General disorders) | 2
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 4
Thyroid function, low (Endocrine disorders) | 1
Anorexia (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Febrile neutrophenia (Blood and lymphatic system disorders) | 2
Infection (Blood and lymphatic system disorders) | 1
Alkaline phosphatase (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
hypophosphatemia (Metabolism and nutrition disorders) | 1
Cognitive disturbance (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Watering Eyes (Eye disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 1
Headache (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes